CLINICAL TRIAL: NCT00302003
Title: A Phase III Study for the Treatment of Children and Adolescents With Newly Diagnosed Low Risk Hodgkin Disease
Brief Title: Combination Chemotherapy Followed by Radiation Therapy in Treating Young Patients With Newly Diagnosed Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHOD0431; NCI-2009-00377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000459962 (Other: Clinical Trials.gov); U10CA098543 (NIH); COG-AHOD0431 (Other: Children's Oncology Group)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2016-08

CONDITIONS: Childhood Favorable Prognosis Hodgkin Lymphoma; Childhood Lymphocyte Depletion Hodgkin Lymphoma; Childhood Mixed Cellularity Hodgkin Lymphoma; Childhood Nodular Sclerosis Hodgkin Lymphoma; Stage I Childhood Hodgkin Lymphoma; Stage II Childhood Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Radiotherapy; Radiation; Doxorubicin; Vincristine; Prednisone; Cyclophosphamide; Ifosfamide; indolepropanol phosphate; Vinorelbine; Dexamethasone; Calcium Dobesilate; etoposide phosphate; Cisplatin; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxorubicin, Vincristine, Cyclophosphamide and Filgrastim (Experimental): Treatment consists of 3 cycles of Doxorubicin hydrochloride IV (25 mg/m2) days 1 & 2, Vincristine sulfate IV (1.4 mg/m2 [max 2.8 mg]) Days 1 & 8, Prednisone orally (40 mg/m2) Days 1-7, Cyclophosphamide IV (600 mg/m2) Days 1 & 2, Filgrastim by mouth or IV (5 micrograms/kg/dose) 24 hours after Cyclophosphamide complete. See detailed description for remainder of therapy.
  Interventions: Radiation: radiation therapy; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Drug: cyclophosphamide; Drug: ifosfamide; Drug: vinorelbine tartrate; Drug: dexamethasone; Drug: etoposide phosphate; Drug: cisplatin; Drug: cytarabine; Biological: filgrastim

INTERVENTIONS:
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Drug: dexamethasone — Given IV
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: etoposide phosphate — Given IV
  Other Names: ETOP; Etopophos
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Biological: filgrastim — Given IV or subcutaneously
  Other Names: G-CSF; Neupogen

SUMMARY:
This phase III trial is studying how well combination chemotherapy works when given before radiation therapy and/or additional chemotherapy in treating young patients with newly diagnosed Hodgkin's lymphoma. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Giving more than one drug (combination chemotherapy) and giving them together with radiation therapy may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Investigate the paradigm of response-based therapy for low-risk Hodgkin's lymphoma by eliminating involved-field radiotherapy (IFRT) in patients who achieve a complete remission (CR) after initial chemotherapy.

II. Investigate whether 3 courses of doxorubicin hydrochloride, vincristine, prednisone, and cyclophosphamide (AV-PC) for the treatment of low-risk Hodgkin's lymphoma is sufficient to induce CR in at least 80% of patients.

III. Investigate whether patients who experience a low-risk relapse after initial treatment with chemotherapy alone can be successfully treated with a salvage regimen comprising ifosfamide and vinorelbine ditartrate with dexamethasone, etoposide phosphate, cisplatin, and cytarabine (IV/DECA) and IFRT.

IV. Maintain the overall survival for patients with low-risk Hodgkin's lymphoma at or above 97%.

V. Determine the prognostic significance of very early response as measured by fludeoxyglucose-positron emission tomography (FDG-PET) or gallium after the first course of chemotherapy.

VI. Evaluate the prognostic significance of elevation of erythrocyte sedimentation rate and C-reactive protein at the time of diagnosis in patients with low-risk Hodgkin's lymphoma on CR rate and relapse rate after chemotherapy alone.

VII. Determine the frequency and severity of late effects of therapy, including thyroid dysfunction, infertility, cardiotoxicity, and second malignant neoplasms.

OUTLINE: This is a multicenter study.

INITIAL CHEMOTHERAPY: Patients receive doxorubicin hydrochloride intravenously (IV) over 10-30 minutes and cyclophosphamide IV over 1 hour on days 1-2, vincristine IV on days 1 and 8, prednisone orally (PO) on days 1-7, and filgrastim (G-CSF) subcutaneously (SC) on days 3-7 and 9-14. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving complete remission (CR) proceed to observation. Patients achieving partial remission proceed to radiotherapy. Patients who have a low-risk relapse after achieving CR on initial chemotherapy proceed to salvage chemotherapy followed by radiotherapy. Patients who have stable disease or disease progression go off study.

SALVAGE CHEMOTHERAPY: Patients receive ifosfamide IV continuously on days 1-4, vinorelbine ditartrate IV over 6-10 minutes on days 1-5, and G-CSF SC or IV beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses. Patients then receive dexamethasone IV over 15 minutes every 12 hours, etoposide phosphate IV over 3 hours every 12 hours, and cytarabine IV over 3 hours every 12 hours on days 1 and 2; cisplatin IV over 6 hours on day 1; and G-CSF SC or IV beginning on day 3 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses. Patients then proceed to radiotherapy.

INVOLVED-FIELD RADIOTHERAPY (IFRT): Beginning 4 weeks after completion of chemotherapy, patients undergo IFRT once daily, 5 days a week, for 2.8 weeks. Patients who do not achieve CR go off study.

After completion of study treatment, patients are followed periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin's lymphoma meeting the following criteria:

  * Newly diagnosed disease
  * Stage IA OR stage IIA without bulky disease
  * No lymphocyte-predominant histology
* Staging on this study will be determined by the clinical stage; surgical staging is strongly discouraged, except for the rare situation of equivocal imaging studies below the diaphragm
* Patients may not have received any previous chemotherapy or radiation therapy; patients may not have received systemic corticosteroids within 30 days of enrollment on this protocol; steroids used for treatment of contrast agent allergy required for computed tomography (CT) scans are acceptable
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^3
* Total bilirubin =< 1.5 x normal
* Alanine (ALT) =< 2.5 x normal
* Shortening fraction >= 27% by echocardiogram OR ejection fraction >= 50% by multi-gated acquisition (MUGA)
* No pathologic prolongation of QTc interval on 12-lead electrocardiography (ECG)
* Female patients of childbearing potential must have a negative pregnancy test
* Lactating females must agree that they will not breastfeed a child while on this study
* Fertile patients must use effective contraception
* Males and females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 287 (Actual)
Dates: Start 2006-02; Primary Completion 2012-03 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Keller, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- [Derived] Parekh A, Keller FG, McCarten KM, Kessel S, Cho S, Pei Q, Wu Y, Castellino SM, Constine LS, Schwartz CL, Hodgson D, Kelly KM, Hoppe BS. Targeted radiotherapy for early-stage, low-risk pediatric Hodgkin lymphoma slow early responders: a COG AHOD0431 analysis. Blood. 2022 Sep 8;140(10):1086-1093. doi: 10.1182/blood.2022016098. PMID 35763667
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxorubicin, Vincristine, Cyclophosphamide and Filgrastim
Started | 287
Completed | 207
Not Completed | 80
Not completed — Lack of Efficacy | 62
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 5
Not completed — Ineligible | 9
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Doxorubicin, Vincristine, Cyclophosphamide and Filgrastim
Number analyzed (Participants) | 287
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 272
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 15 [3 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 227
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 220
  More than one race | 0
  Unknown or Not Reported | 27
Region of Enrollment [Number; unit: participants]
  United States | 250
  Australia | 3
  Canada | 25
  Israel | 1
  Mexico | 1
  New Zealand | 2
  Puerto Rico | 4
  Switzerland | 1

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival Without Receiving Radiation Therapy (EFSnoRT).
Description: Survival is defined as the minimum time from study entry to requirement for additional chemotherapy and IFRT for retrieval, occurrence of a second malignant neoplasm, or death from any cause. Patients without report of such events where censored at last contact. Patients who achieve less than CR after 3 cycles of AV-PC will require IFRT and hence will satisfy this definition at the time of response evaluation. Patients who achieve a CR but who relapse will receive addition chemotherapy and IFRT or intense retrieval and hence will satisfy this definition at the time of the first relapse of Hodgkin disease. This endpoint will be used to compute event free survival without receiving radiation therapy (EFSnoRT).
Time Frame: At 60 months
Population: Eligible (n=278) and evaluable response and review of response, n=275. Follow-up for censored patients (n=138) is 76 months (range: 1.8 to 108 months).
Measure: Number (95% Confidence Interval); unit: Probability of survival
Groups:
- Group 1: Doxorubicin, Vincristine, Cyclophosphamide and Filgrastim
Arm/Group | Group 1
Number analyzed (Participants) | 275
Probability of survival | 0.49 [0.42 to 0.54]

2. Primary Outcome: Intensive Therapy Free Survival (ITFS).
Description: Survival is defined as the minimum time from study entry to a relapse of higher risk at any time, any relapse following treatment with protocol mandated IFRT, death from any cause, or the occurrence of a second malignant neoplasm. This will be used to compute intensive therapy free survival (ITFS). Patients without report of such events where censored at last contact. This differs from traditional EFS in that relapse after AVPC* x3 therapy alone that does not place the patient in a higher risk category is not considered a treatment failure. In this definition, higher-risk relapse refers to relapse involving sites and extent of disease that place the patient in the current COG definition of intermediate or high-risk disease. If a patient with CR who experiences a LR relapse is not retreated with protocol-mandated chemotherapy and IFRT, subsequent disease relapses will nevertheless be counted in the analysis of the treatment strategy.
Time Frame: At 60 months
Population: Eligible (n=278) and evaluable response and review of response, n=275. Follow-up for censored patients (n=245) is 76 months (range: 4.7 to 109 months).
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Group 1
Number analyzed (Participants) | 275
Probability of survival | 0.89 [0.84 to 0.92]

3. Primary Outcome: Event Free Survival (EFS)
Description: Survival is defined as the minimum time from study entry to a relapse of any kind, death from any cause, or occurrence of a second malignant neoplasm. Patients without report of such events where censored at last contact. This will be used to compute event free survival (EFS).
Time Frame: At 60 months
Population: Eligible (n=278). Follow-up for censored patients (n=223) is 75 months (range: 4.7 to 108 months).
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Group 1
Number analyzed (Participants) | 278
Probability of survival | 0.79 [0.74 to 0.84]

4. Secondary Outcome: Overall Survival
Description: Survival is defined as time from study entry to death due to any cause. Patients alive at last contact where censored at last contact.
Time Frame: At 60 months
Population: Eligible (n=278). Follow-up for censored patients (n=277) is 76 months (range: 4.7 to 109 months).
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Group 1
Number analyzed (Participants) | 278
Probability of survival | 0.99 [0.97 to 1.00]

ADVERSE EVENTS:
Arm/Group | Doxorubicin, Vincristine, Cyclophosphamide and Filgrastim
Serious Adverse Events (participants affected / at risk) | 2/278
Other Adverse Events (participants affected / at risk) | 80/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin, Vincristine, Cyclophosphamide and Filgrastim (N=278)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
CPK increased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin, Vincristine, Cyclophosphamide and Filgrastim (N=278)
Febrile neutropenia (Blood and lymphatic system disorders) | 18 (18)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Delayed puberty (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (10)
Oral pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (10)
Fatigue (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 12 (12)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 4 (4)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (7)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Neuralgia (Nervous system disorders) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.